CLINICAL TRIAL: NCT05521464
Title: Robert Jones Bandage Versus Cast in the Treatment of Distal Radius Fracture in Children: a Randomized Controlled Trial
Brief Title: Robert Jones Bandage Versus Cast in the Treatment of Distal Radius Fracture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Jagar Omar Doski, Assistant Professor of orthopedics, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jagar Omar
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Fracture Distal Radius; Children, Only
Keywords: Robert Jones bandage; cast
MeSH Terms: conditions — Wrist Fractures | interventions — POLR1G protein, human; Calcium Sulfate

STUDY DESIGN:
Intervention Model Description: randomized controlled non-inferiority clinical trial of patients based on a parallel-group type with an allocation ratio of 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Cast by Plaster of Paris
  Interventions: Other: cast
- Group 2 (Experimental): Robert Jones bandage
  Interventions: Other: Robert Jones Bandage

INTERVENTIONS:
Other: cast — Application of a short arm cast from just below the elbow to the finger's knuckles. The cast was from a Plaster of Paris bandage over a cotton pad. The participants who received this treatment modality were considered group 1 (control group)
  Other Names: Plaster of Paris
  Arms: Group 1
Other: Robert Jones Bandage — Modified RJ bandage (firmly applied two layers of bulky cotton layers alternating with two layers of elastic bandage in the following order: bandage - cotton - bandage - cotton - bandage). It was applied from below the elbow to the finger's knuckles. The participants who received this treatment modality were considered group 2 (trial group).
  Other Names: Crepe bandages plus cotton rolls
  Arms: Group 2

SUMMARY:
Aim and objectives This study aimed to treat fractures of the distal end of the radius in the children with Robert Jones (RJ) bandage in comparison with a cast. The objective was to compare the frequency of occurrence of the complications, child comfortability, and family satisfaction with this treatment modality.

DETAILED DESCRIPTION:
Methods Study type and approvals The study was a randomized controlled non-inferiority clinical trial of patients based on a parallel-group type with an allocation ratio of 1:1.

Sittings The study was done in the emergency reception unit and the orthopedic unit of Duhok Emergency Teaching Hospital (single-center study), Duhok city, Iraq during the period extending from October 2021 to August 2022.

The study was conducted by a team from the hospital composed of a consultant Orthopedic surgeon (person 1), a permanent resident orthopedic doctor (person 2), and a radiologist (person 3). Person 1 generates the random allocation sequence, assessed the outcome clinically, analyzed the results, and drafted the article. Person 2 enrolled the participants in the study, assigned the interventions, and drafted the article. Person 3 assessed the outcome radiologically.

Interventions The participants included received one of the modalities of treatment planned for this study. The first modality was by application of a short arm cast from just below the elbow to the finger's knuckles. The cast was from a Plaster of Paris bandage over a cotton pad. The participants received this modality of treatment considered as group 1 (control group). The second modality was the modified RJ bandage (firmly applied two layers of bulky cotton layers alternating with three layers of elastic bandage in the following order: bandage - cotton - bandage - cotton - bandage)[17]. It was applied from below the elbow to the finger's knuckles. The participants received this modality of treatment considered as group 2 (trial group).

The participants and their companions were instructed to keep their modality of treatment clean and dry. Both groups asked for frequent follow-up (at the end of the 2nd, 4th, 6th, and 12th week) until the fracture unit. At each follow-up visit, the participant was checked for possible complications. The final assessment was done at the end of the 12th week by the consultant orthopedic doctor in collaboration with the radiologist.

Sample size calculation The assumed sample size was calculated by using the G*Power 3.1.9.7 computer software program. A minimum of 148 participants (74 for each group) was required to have a power of 80% chance of detecting the difference between the groups, and a two-sided 95% level of confidence (0.05 level of significance) to avoid the type 1 -alpha- error, with a probable hypothetical effect size of about 0.3 and a degree of freedom of 1 in the contiguity table.

Randomization The allocation of the participants into the modalities of the treatment was done by a simple randomization method with an allocation ratio of 1:1. It was generated by using the website program www.randomization.com. The first generator of the program was used to randomize 148 subjects into both modalities of treatment blocks (74 casts, 74 RJ bandages) (seed 7180). The random allocation sequence was generated by person 1 from the team of the study. It was concealed from the rest of the study team. Person 2 enrolled the participants in the study (assessed the eligibility of the cases, obtained the informed consent) and assigned the interventions.

Blinding The team of the study (apart from person 3 - the radiologist) was not blinded to the modality of treatment that they provided to the patients. The radiologist who assessed the radiological outcome of the cases was blinded to the modalities of treatment. The participants were blinded to the result of the treatment of the other patients included in this study.

The data collection

The data was collected in a special paper for each patient separately. The data included were divided into two parts:

Part 1 included the basic demographic data of the patient and injury like name, age, gender, place of living, date of a wrist injury, type of wrist injury (proved by the radiographic film), type of treatment (group), the time interval between the injury and beginning of treatment, duration of treatment, dates of each follow up. Part 2 included the outcomes during each follow-up visit and at the final assessment like complications of treatment, patient comfortability, and family satisfaction.

Statistical analysis The data analysis was done by admitting the collected data into the Statistical Package for Social Sciences (SPSS) software computer program (IBM Corp. Released 2015. IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp.). The statistical analysis included the standard descriptive statistics used to describe the basic descriptive data of the patients and injuries. The means and standard deviations (SD) or medians and interquartile ranges were used for the continuous variables, while frequencies and percentages were used for the categorical variables. The comparison between the outcomes of the treatment modalities in both groups was done by finding the difference between the summary statistics in the chi-squared test. The difference was considered statistically significant when the p-value was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 2-12 years old age.
* Sex: both male and female.
* Duration of symptoms: less than 5 days.
* Type of injury: fracture at the distal end of radius proofed by a radiograph film in two views (posteroanterior and lateral).
* Type of fracture: the fracture which is usually treated conservatively -without intervention- like:

  1. torus (buckle) metaphyseal fracture
  2. greenstick fracture
  3. undisplaced or minimal displaced fracture distal radial physis (Salter-Harris classification type 1 and 2 only) that does not need reduction
  4. undisplaced or minimal displaced metaphyseal fracture that doesn't need reduction (a tilt of fewer than 15 degrees and shift less than 5 millimeters at the fracture site in both views).

Exclusion Criteria:

* open fractures
* pathological fractures
* displaced fractures that need reduction
* delayed presentation beyond five days
* associated fracture of the ulnar bone
* polytraumatic cases.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Number of complications | 6-12 weeks
  The complications were considered to be present if one of the following was noticed:
  1. Skin problems like pressure soreness, skin irritation, itching, and dermatitis.
  2. Bone deformity due to a displacement of the bone fragments at the fracture site to an unacceptable degree (tilt more than 15 degrees and/or shift more than 50% of the bone width at the fracture site) confirmed by the report of the radiologist, or due to growth disturbance from growth plate damage.
  3. Joint stiffness by limitation of the wrist movements (limitation of more than 10 degrees in any direction).
  4. Refracture within 12 weeks.

SECONDARY OUTCOMES:
Child comfortability with the treatment modality. | 6 weeks
  yes or no
Family satisfaction the treatment modality. | 6-12 weeks
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Jagar O Doski, Ph.D., Principal Investigator — College of Medicine, University of Duhok, Duhok, Iraq.
Locations (1):
- Jagar Omar Doski, Duhok, Duhok Governorate / Kurdistan Region, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Data will be provided by the authors on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: directly after publication of the article and whenever requested.
Access Criteria: email: jagaromar@uod.ac

REFERENCES:
- [Background] Hedstrom EM, Svensson O, Bergstrom U, Michno P. Epidemiology of fractures in children and adolescents. Acta Orthop. 2010 Feb;81(1):148-53. doi: 10.3109/17453671003628780. PMID 20175744
- [Background] Wilkins KE. Principles of fracture remodeling in children. Injury. 2005 Feb;36 Suppl 1:A3-11. doi: 10.1016/j.injury.2004.12.007. PMID 15652934
- [Background] Al-Ansari K, Howard A, Seeto B, Yoo S, Zaki S, Boutis K. Minimally angulated pediatric wrist fractures: is immobilization without manipulation enough? CJEM. 2007 Jan;9(1):9-15. doi: 10.1017/s1481803500014676. PMID 17391594
- [Background] Do TT, Strub WM, Foad SL, Mehlman CT, Crawford AH. Reduction versus remodeling in pediatric distal forearm fractures: a preliminary cost analysis. J Pediatr Orthop B. 2003 Mar;12(2):109-15. doi: 10.1097/01.bpb.0000043725.21564.7b. PMID 12584495
- [Background] Edmonds EW. No difference in improvement in physical function between splint and cast at 6 weeks in children with minimally angulated fractures of the distal radius. Evid Based Med. 2011 Apr;16(2):49-50. doi: 10.1136/ebm1161. Epub 2010 Dec 7. No abstract available. PMID 21139033